CLINICAL TRIAL: NCT06839976
Title: CD19-Directed Chimeric Antigen Receptor Autologous T Cells (CART19) for Adolescents and Young Adults With Systemic Lupus Erythematosus (SLE)
Brief Title: CD19-Directed Chimeric Antigen Receptor Autologous T Cells (CART19) for Lupus
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-022668
Record Dates: First submitted 2025-02-12; First posted 2025-02-21 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: SLE; Systemic Lupus Erythematosus (SLE); CAR T Cell; CART19; Cell Therapy; Lupus; Lupus Nephritis (LN)
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis | interventions — CTL019 chimeric antigen receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CART19 (Experimental): Participants will receive the study product. CART19 cells transduced with a lentiviral vector to express anti-CD19 scFv:41-BB:TCRζ, administered by IV injection.
  Interventions: Biological: CART19

INTERVENTIONS:
Biological: CART19 — CART19 cells transduced with a lentiviral vector to express anti-CD19 scFv:41-BB:TCRζ, administered by IV injection.

SUMMARY:
This is a single-center, single-arm, open-label phase 1/2 study of CART19 in children and young adults with refractory Systemic lupus erythematosus (SLE), including both patients diagnosed with lupus nephritis (LN) and patients with non-renal Systemic lupus erythematosus (SLE).

Phase 1 will evaluate the safety of CART19 in 6-12 patients with Systemic lupus erythematosus (SLE). There is no planned dose escalation, but a dose de-escalation will be made based on the incidence of Dose Limiting Toxicities. Phase 2 will evaluate the efficacy and further evaluate the safety of CART19 in this population.

DETAILED DESCRIPTION:
Lupus disease activity is associated with increased numbers of activated naïve B cells and polyclonal expansion of antibody secreting cells, indicating a central role for B cells in the pathogenesis of SLE. While traditional anti-CD19 antibody therapies have been utilized with varying success in the treatment of Systemic lupus erythematosus (SLE), CD19 directed cellular therapies have emerged as an attractive therapeutic option that may lead to immunosuppression-free remission in this population given the ability of CD19 directed CAR T cells to more deeply deplete the B cell compartment. Previous clinical experience utilizing CD19 directed CAR T cells in patients diagnosed with Systemic lupus erythematosus (SLE) have exceeded any other Systemic lupus erythematosus (SLE) therapeutic available; although, those clinical trials have treated a limited number of subjects. During this trial the test article will be CART19 cells transduced with a lentiviral vector to express anti-CD19 scFv:41-BB:TCRζ, administered by IV injection.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form must be obtained prior to any study procedure. Labs or other procedures obtained during routine clinical care may be used for eligibility if obtained within the protocol required window.
2. Patient age must be 12-29 years, inclusive, at time of enrollment.
3. Meeting ACR/EULAR Classification Criteria for SLE
4. ANA positive > 1:80 and/or double-stranded DNA (dsDNA) positive
5. Active (refractory) disease, despite at least three months of conventional therapy, defined as follows:

   a. Lupus nephritis subjects must meet both the following criteria: i. ISN/RPS active nephritis Class III/IV +/- V lupus nephritis diagnosed by biopsy within past 12 months.

ii. Persistent and clinically significant: ≥2 measurements with urine protein on first morning sample with either of the following:

1. > 1000mg/g creatinine
2. > 500 mg/g creatinine associated with renal dysfunction or low albumin.
3. > 500 mg/g creatinine in a patient with rising proteinuria after prior complete renal response b. Non-renal SLE subjects must meet either of the following criteria: i. SLEDAI-2K ≥ 8 and clinical SLEDAI-2K ≥ 6 ii. Inability to decrease prednisone ≤7.5mg/day or 0.15mg/kg/day, whichever is lower, due to active disease.

6. Patients must have had at least 3 months conventional therapy defined as:

1. Conventional induction immunosuppressive agent(s) (mycophenolate mofetil or cyclophosphamide), and
2. At least one additional therapy:

i. B-cell directed biologic therapy (e.g., rituximab, belimumab, ofatumumab, obinutuzumab) ii. Calcineurin inhibitor (e.g., tacrolimus, cyclosporine, voclosporin) iii. Other immunosuppressive medication for SLE (e.g., anifrolumab, abatacept, JAK inhibitor, others) 7. Adequate organ function status

1. Renal: eGFR must be ≥30 and subject cannot be receiving dialysis.
2. Hepatic: Transaminases < 5x upper limit of normal and serum conjugated (Direct) bilirubin <1.5x upper limit of normal unless attributable to SLE. If attributable to autoimmune disease, Child-Pugh score must be class A or class B. Child-Pugh score cannot be class C.
3. Cardiac: Shortening fraction > 28%, left ventricular ejection fraction >45%, and no evidence of severe pulmonary hypertension
4. Pulmonary: Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and <Grade 3 hypoxia; DLCO ≥40% (corrected for anemia and/or VA volume) if PFTs are clinically appropriate as determined by the treating investigator.

   8. Subjects of reproductive potential must agree to use acceptable birth control methods.

Exclusion Criteria:

1. Active, untreated infections
2. HIV infection
3. Active Hepatitis B

   a. Patients must have a negative hepatitis B surface antigen to be enrolled on this study.
4. Active Hepatitis C
5. Patients with severe neuropsychiatric lupus or neurologic manifestations of SLE (e.g. stroke, seizure, psychosis, demyelinating syndromes, organic brain syndrome, or lupus related headaches)
6. Monogenic lupus (known)
7. Previous autologous or allogenic stem cell transplant
8. Previous kidney transplant
9. History of seizure disorder
10. Patients who are on anti-epileptic therapy
11. Participation in a clinical trial in which the patient receives an investigational drug within a time period equal or less than 5.5 half-lives of the investigational agent prior to study enrollment.
12. Subjects who are unwilling or unable to discontinue immunosuppressive medications at the times of T cell collection and CART19 infusion
13. Any comorbidity that in the opinion of the investigators would jeopardize the ability of the subject to tolerate therapy.
14. Pregnant patients. All participants of childbearing potential must have negative pregnancy test.
15. Lactating participants who want to continue breastfeeding.
16. Patients who are unwilling to consent to LTFU

Ages: 12 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Frequency of the dose limiting toxicities of CART19 | up to 24 months post infusion
  Frequency of the dose limiting toxicities of CART19

SECONDARY OUTCOMES:
Rate of childhood SLE Clinical Remission off steroids (cCR-0) at 3 months | 3 months post treatment
2-year overall survival rate | 24 months post infusion
2-year flare free survival rate | up to 24 months post infusion
Feasibility of manufacturing CART19 for participants with SLE | up to 24 months post infusion
  Feasibility of manufacturing CART19 measured by the percentage of manufactured products that do not meet release criteria for vector transduction efficiency, T cell product purity, viability, or sterility
Proportion of patients achieving a complete renal response | up to 24 months post infusion
  renal response will be measured by urine protein/creatinine ratio of < 0.5, normal renal function (serum creatinine ≤ULN) without worsening of baseline serum creatinine by more than 15%, and inactive urinary sediment (<10 red blood cells (RBCs)/high-power field (HPF) without RBC casts)
Proportion of patients achieving a partial renal response | up to 24 months post infusion
  partial renal response will be measured by urine protein/creatinine ratio of < 0.5, normal renal function (serum creatinine ≤ULN) without worsening of baseline serum creatinine by more than 15%, and inactive urinary sediment (<10 red blood cells (RBCs)/high-power field (HPF) without RBC casts)
Rate of CART19 expansion, persistence or B cell aplasia | up to 24 months post infusion
  Rate of CART19 expansion, persistence and B cell aplasia will be measured by qPCR and flow cytometry
Survival of CART19 cells | up to 24 months post infusion
  CART19 cell survival will be measured by utilizing polymerase chain reaction analysis of whole blood to detect and quantify number of cells over time.
Elevations in cytokines in serum | up to 24 months post infusion
  to assess bioreactivity and biological response following CART cell infusion, systemic soluble immune and inflammatory factors will be measured by assessing any change in elevations in cytokines in serum prior to infusion and after.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Elgarten, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No